CLINICAL TRIAL: NCT00154583
Title: Comparison of the Human Papillomavirus (HPV) Type 16 E7-Specific Immune Response Between a Normal Population and Patients With Cervical Lesions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9261701445
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2006-12-21 (Estimated); Status verified 2003-01

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; human papillomavirus; cancer vaccine; normal volunteer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Cervical cancer is the most frequent neoplasm and the third in mortality rate of the malignancies in women in the world. It results in about 200,000 women dying of cervical cancer each year worldwide. The available forms of treatment - surgery, radiation therapy, and chemotherapy - are all cytoreductive treatment modalities, so, in addition to killing cancerous cells, healthy cells are also destroyed in the process. Indeed, there is a need to decrease the incidence of cervical cancer and develop better forms for its treatment.

Human papillomaviruses (HPV) have been consistently implicated in causing cervical cancer especially those high-risk types (HPV 16, 18, 31, 45) which have been strongly associated with cervical cancer. HPV 16 was found in more than 50% of cervical cancer tissues. So, the host immune response plays an important role in determining the regression of a cervical abnormality or persistence and progression to a malignancy via targeting HPV.

The ideal cancer treatment should be able to eradicate systemic tumors at multiple sites in the body while having the specificity to discriminate between neoplastic and nonneoplastic cells. In this regard, antigen-specific cancer immunotherapy represents an attractive approach for cancer treatment. By cooperating with Dr. TC Wu at the Johns Hopkins Medical Institutes, the investigators have recently developed some E7-specific cancer vaccines of different strategies such as DNA, or replication-defective SINrep5 virus. They found that these E7-chimeric DNA vaccines are capable of preventing and treating the growth of murine model tumors expressing E7. These positive results from the preclinical murine models have encouraged the investigators to focus on the development of a cancer vaccine and immunotherapy and apply these vaccines to human subjects. However, it is very important to set up various E7-specific immunologic assays of human beings to evaluate the effects of a cancer vaccine or immunotherapy in future clinical trials. So the investigators would like to provide this proposal to address the development of HPV 16 E7-specific immunologic assays in human beings. There are two main goals in this study. First, the investigators would like to establish and compare the differences of HPV type 16 E7-specific immunologic responses between the normal population, people with HPV infection, patients with cervical intraepithelial neoplastic (CIN) lesions, and patients with cervical cancer. Second, they would like to correlate the disease severity of cervical cancer with the immunologic responses to HPV type 16 E7 antigen.

DETAILED DESCRIPTION:
HPV and Cervical Cancers:

Human papillomaviruses (HPV) are small, nonenveloped DNA viruses which induce epithelial tumors of skin or mucosa. The majority of tumors are benign, show limited growth and usually regress spontaneously. However, a number of human papillomaviruses induce tumors that may eventually progress to carcinomas. The genital HPV types 16 and 18, and less frequently, types 31, 33, 35, 45, 51 and 56, have been implicated in the etiology of cervical and other anogenital cancers. Approximately 500,000 women worldwide develop cervical cancer yearly and it is the second leading cause of death from cancer in women. In developed countries, cancer of the cervix ranks behind cancers of the breast, lung, uterus, and ovaries and accounts for 7% of all female cancers. In the United States, there are about 4,800 deaths annually from cervical cancer. The evidence linking HPVs to anogenital cancer comes from epidemiologic and laboratory studies. More than 90% of cervical cancers and their precursors, so-called cervical intraepithelial neoplasia (CIN), contain human papillomavirus (HPV) DNA sequences. The HPV types found in cancer cells have transforming activity in in vitro studies and the viral transforming proteins, E6 and E7, are consistently expressed in cervical cancer cell lines and in HPV-associated cancers of patients. In HPV-associated malignant transformation, viral DNA may be integrated into the cellular DNA and integration often results in deletion of large sectors of the viral genome. Late genes (L1 and L2) and some early genes (E1 and E2) are usually lost, leaving E6 and E7 as the only open reading frames frequently found in carcinomas. Expression of E6 and E7 is likely to overcome the regulation of cell proliferation normally mediated by proteins like p53 and Rb, allowing uncontrolled growth and providing the potential for malignant transformation.

HPV Oncogenic Proteins, E6 and E7, as Ideal Targets for the Development of Antigen-Specific Immunotherapies or Vaccines for HPV-Associated Cervical Malignancies:

E6 and E7 represent ideal targets for the development of antigen-specific immunotherapies or vaccines for HPV-associated malignancies. First, more than 90% of cervical cancers have been associated with HPVs, particularly type 16, and E6 and E7 are consistently expressed in most cervical cancers. Second, while most tumor specific antigens are derived from normal proteins or mutated proteins, E6 and E7 are completely foreign viral proteins, and potentially may harbor more antigenic peptides/epitopes than a mutant protein (i.e. p53) or a reactivated embryonic protein (i.e. MAGE-1). Third, since E6 and E7 are required for the induction and maintenance of malignant phenotypes of cancer cells, cells of cervical cancer cannot evade an immune response through antigen loss. Without functional E6 and E7, these cells would cease to be tumorigenic. Therefore, E6 and E7 proteins represent ideal targets for developing antigen-specific immunotherapies or vaccines for cervical cancer.

Various forms of vaccines, such as vector-based vaccines, tumor-based vaccines, DNA based vaccines and protein/peptide-based vaccines have been described in experimental systems targeting HPV-16 E6 and/or E7 proteins. For example, Meneguzzi et al. reported that inoculation of rats with vaccinia recombinants expressing HPV-16 E6 or E7 retarded or prevented tumor development in 25-47% of rats challenged with a tumorigenic rat cell line co-transfected with HPV-16 and activated ras. In addition, Chen et al. demonstrated that immunization of mice with syngeneic non-tumorigenic cells transfected with the HPV-16 E7 gene confers protection against transplanted HPV-16 E7 positive syngeneic tumor cells. Feltkamp et al. identified a CTL epitope in HPV-16 E7 using H-2Kb and H-2Db MHC class I-peptide-binding studies. Immunization with this peptide rendered mice resistant to a challenge with HPV-16 transformed tumor cells. Furthermore, chimeric papillomavirus-like particles (CVLPs) consist of HPV-16 L1-E7 (Nieland et al., personal communication) or HPV-16 L1/L2-E7 (Greenstone et al., personal communication) chimeric proteins have been used as therapeutic vaccines against HPV-16 E7 expressing tumors in murine models. More recently, a phase I/II clinical trial was performed in eight patients with late stage cervical cancer using a live recombinant vaccinia virus expressing the E6 and E7 proteins of HPV 16 and 18 (TA-HPV). In that study, no significant clinical side-effects or environmental contamination by live TA-HPV were observed.

Importance of Cell Mediated Immune Responses in Controlling both HPV Infections and HPV-Associated Neoplasms:

Several lines of evidence suggest that cell mediated immune responses are important in controlling both HPV infections and HPV-associated neoplasms. First, the prevalence of HPV-related diseases (infections and neoplasms) is increased in transplant recipients and human immunodeficiency virus (HIV) infected patients, both of whom are known to have impaired cell mediated immunity. Second, animal studies have demonstrated that immunized animals are protected from papillomavirus infection and from the development of neoplasia. Immunization also facilitates the regression of existing lesions. Third, infiltrating CD4+ (T helper cells) and CD8+ (cytotoxic/suppressor T cells) T cells have been observed in spontaneously regressing warts and fourth, warts in patients who are on immunosuppressive therapy often disappear when this treatment is discontinued.

Cellular Immune Responses to HPV:

The understanding of T-cell mediated immunity to HPV infections was facilitated by identification of MHC class I and class II epitopes of HPV proteins. Several groups have attempted to map murine and human T helper (Th) cell epitopes on HPV proteins. Several groups have also tried to map murine as well as human cytotoxic T-lymphocyte (CTL) epitopes on HPV proteins. Kast et al. have identified several high affinity binding peptides of HPV-16 E6 and E7 proteins for human HLA-A alleles. Furthermore, HPV-specific CTLs recognizing HPV E6 and E7 proteins have been demonstrated in peripheral blood of cervical cancer patients, in healthy donors and in patients with CIN lesions [Nakagawa, 1997 #562]. Furthermore, infiltration of cervical cancer tissue with HPV-specific CTLs has been recently described.

Cell-mediated immune responses in HPV-infected lesions can be demonstrated by in vivo skin tests, in vitro CTL assays and in vitro lymphoproliferative responses. For instance, Hopfl et al. have used bacterially-expressed HPV-16 proteins for skin tests in patients with CIN lesions and have found specific skin responses to the virion protein L1 and not the E4 protein. In patients with CIN lesions, HPV-specific CTLs have been identified in PBMC and in cervical tissues. The in vitro lymphoproliferative responses in patients with CIN lesions have been actively investigated. For example, de Gruijl et al. reported that T cell proliferative responses against HPV-16 E7 oncogenic protein were most prominent in CIN patients with a persistent HPV infection. However, Kadish et al. reported that lymphoproliferative responses to specific HPV-16 E6 and E7 peptides appeared to be associated with the clearance of HPV infection and the regression of CIN lesions.

Importance of Helper T Cell Functions in Generating Effective Antitumor Responses:

Increasing evidence has suggested that inadequate antitumor responses can result from a failure of the helper arm of the immune response. The events leading to the activation of CTL are tightly regulated in order to protect against the development of inappropriate immune responses to self antigens or exaggerated responses to foreign antigens. This regulation is mediated by lymphokines produced by CD4+ T helper cells. CD4+ T helper cells are critical to the generation of potent antitumor immune responses. CD4+ T cells have been shown to be instrumental in generating immune responses against several solid malignancies in murine [Fearon, 1990 #833; Golumbek, 1991 #834] and in human populations [Topalian, 1994 #396; Topalian, 1994 #397]. Several mouse tumors that are transfected with syngeneic MHC class II genes become very effective vaccines against subsequent challenge with wild type class II negative tumors [Ostrand-Rosenberg, 1990 #177; James, 1991 #272; Chen, 1993 #213] In addition, as crucial memory cells in the T cell arm of the immune system, CD4+ cells may be able to provide long term immunity against specific antigens [Tew, 1990 #624; Sprent, 1994 #625].

Role of Cytokines in Cell-Mediated Immunity:

Cell mediated immunity is regulated by cytokines which are secreted by T helper cells. In general, T helper cells can be classified as Th1 and/or Th2 cells based on the different types of cytokines they secrete. Th1 cells secrete interleukin (IL) 2 and interferon gamma (IFN-gamma). Th2 cells produce IL-4, IL-5, IL-10 and IL-13. The Th1 lymphocytes are the most important effector cells in inflammatory reactions associated with vigorous delay-type hypersensitivity but low antibody production, as occurs in contact dermatitis and in viral or intracellular bacterial infections (for review, see [Mosmann, 1989 #168; Romagnani, 1992 #130]). The functional phenotype of most Th2 cells may account for both the persistent production of certain antibody isotypes, particularly IgG1 and IgE, and the eosinophilia observed in human helminthic infections and allergic disorders. Lymphocyte mediated protection from viral infections as well as control of tumors is thought to be mediated by Th1 cytokine responses and impaired by Th2 cytokine responses. The IL-2 and IFN-gamma producing Th1 response is likely to be the major component that contributes to the development of cell mediated immunity against HPV infections and HPV-associated neoplasms.

Chimeric E7-specific vaccines can control the HPV16 E7-expressing tumor model. By cooperating with Prof. TC Wu at the Johns Hopkins Medical Institutes, we have successfully developed several chimeric DNA, RNA, and virus-vector vaccines to prevent and treat HPV16 E7-expressing tumors in animal models. We found that these E7-chimeric DNA vaccines are capable of preventing and treating the growth of murine model tumors expressing E7. These positive results from the preclinical murine models have encouraged us to focus on the development of a cancer vaccine and immunotherapy and apply these vaccines to human subjects.

However, it is very important to set up various E7-specific immunologic assays of human beings to evaluate the effect of a cancer vaccine or immunotherapy in future clinical trials. So we would like to provide this proposal to address the development of HPV 16 E7-specific immunologic assays in human beings. There are several aims in this project:

1. to develop and utilize assays to measure CTLs to HPV 16 E7 proteins, and
2. to develop and utilize assays to measure T helper (Th) responses to HPV 16 E7 antigens.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* People infected with HPV type 16 but without CIN lesions
* Patients with CIN lesions
* Patients with cervical cancer from National Taiwan University Hospital
* Informed consent is obtained, and the protocols are reviewed and approved by the appropriate Investigative Review Boards.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2003-01; Study Completion 2008-12

CONTACTS AND LOCATIONS:
Overall Officials: Chi-An Chen, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan